CLINICAL TRIAL: NCT05555537
Title: Role of Plasma miRNA223 and High Mobility Group Box 1(HMGB1) as Predictors of Drug Resistant Epilepsy
Brief Title: MiRNA223 and HMGB1 as Apredictos for Drug Resistant Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Ali Samir Hussien Mohamed, Assistant lecture, Assiut University
Other Study IDs: drug resistant epilepsy
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drug resistant epilepsy: failure to achieve sustained seizure freedom after adequate and well tolerated trials of two antiseizure medications
  Interventions: Diagnostic Test: MiRNA223 and High mobility group box1(HMGB1)
- Medically controled epilepsy: seizure freedom for at least the last 6months) matched in sex and age.
  Interventions: Diagnostic Test: MiRNA223 and High mobility group box1(HMGB1)

INTERVENTIONS:
Diagnostic Test: MiRNA223 and High mobility group box1(HMGB1) — Measure tye 2 biomarkers miRNA223 and HMGB1 in drug resistant and in medically controled epilepsy

SUMMARY:
Evaluation of the role of estimation of serum level of miRNAs223 and HMGB1in detection of patient with drug resistant epilepsy.

Early detection of the prognosis might help in guiding patients for proper management and treatment strategy.

This may open the door for new drug trials.

DETAILED DESCRIPTION:
Epilepsy is the most prevalent neurological disorders (1). Drug-resistant epilepsy (DRE) represent approximately 30% of epilepsy..DRE is defined as failure to achieve sustained seizure freedom after adequate and well tolerated trials of two antiseizure medications( ASMs).The identification of circulating biomarkers for DRE could give an early idea about the prognosis and improve the choice of correct treatment.

MiRNAs are small noncoding RNAs that span between 19 and 24 nucleotide bases((2).They gain biological activity through base pairing in the 30-untranslated regions of target messenger RNA (mRNA) , thereby guiding a protein complex termed the RNA-induced silencing complex (RISC) that bind to the mRNA sequence and results in either the inhibition of translational processes or the degradation of the mRNA (3). Dysregulated miRNA expression has been associated with inflammatory pathways, cell death, neuronal excitability, and synaptic reorganization, which underlie epileptogenesis (4).

High- mobility group box 1(HMGB1) is a chromatin component that is physiologically attached to nuclei. However, following CNS insult, it can promptly be migrated towards cytoplasm and is discharged extracellularly. HMGB1mediates sterile neuro-inflammation evoked by epileptogenic injury and recurrent seizures(5) .HMGB1 increases in neurons, glia, and endothelial cells of the blood brain barrier (BBB) in DRE.

The HMGB1 contributes to the overexpression of P-glycoprotein, a BBB protein, which is induced in DRE foci and extrudes various ASMs from the brain(6) .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as drug resistant epilepsy .
* Control group: patients diagnosed as medically controlled epilepsy

Exclusion Criteria:

* Symptomatic epilepsy (vascular, tumor, post encephalitic, syndromic and febrile seizures).
* Alzheimers disease
* Parkinsons disease
* amyotrophic lateral sclerosis
* major depression disorder
* Non neurological criteria: tumors and cardiovascular

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Drug resistant epilepsy defined as(failure to achieve sustained seizure freedom after adequate and well tolerated trials of two anti-seizure medications) Well controlled epilepsy defined as(seizure freedom for at least the last 6months) matched in sex and age.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
role of estimation of serum level of miRNAs223 and HMGB1in detection of patient with drug resistant epilepsy. | 2year
  Early detection of being drug resistant epilepsy might help in guiding patients for proper management and treatment strategy.